CLINICAL TRIAL: NCT05378958
Title: Qualitative Phenomenological Study on Remote Therapeutic Education by Videoconferencing Crossing the Participant and Caregiver View
Brief Title: Qualitative Phenomenological Study on Videoconferencing Therapeutic Education
Acronym: Visio ETP
Status: Withdrawn | Type: Observational
Why Stopped: Investigators were unable to begin and conduct the research.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220260; 2022-A00093-40 (Other: IDRCB Number)
Record Dates: First submitted 2022-05-02; First posted 2022-05-18 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2024-03

CONDITIONS: Chronic Disease
Keywords: Chronic disease; Therapeutic patient education; Pediatric therapeutic education; Videotherapeutic conferencing education; Understanding videoconferencing therapeutic education through lived experience; Recommendations on videoconferencing therapeutic education; Promotion of videoconferencing therapeutic education
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Caregivers: Any health professional (medical or paramedical profession) practicing therapeutic education in distance mode by videoconferencing, regardless of the programs concerned
  Interventions: Other: Individual interview
- Participants: * Patient's caregivers or parents who have taken part in a therapeutic education session by videoconference (individual or collective) as part of a program, regardless of their age, sex or the pathology concerned by education program
  * Patients: from 10 years old and only if the therapeutic education session was intended for them, regardless of gender or pathology
  Interventions: Other: Individual interview

INTERVENTIONS:
Other: Individual interview — Individual semi-directed explication interview with phenomenological questioning centered on lived experience.
  The individual interview aims to collect data by questioning the participants using interview communication techniques, essentially on the "reformulation" technique. The interview is structured using an interview guide containing the list of open questions with prompts to be answered during the discussion.

SUMMARY:
Therapeutic patient education (TPE) is one of the mechanisms that make patients with chronic disease as competent as possible to manage illness and treatment by helping them to be autonomous and responsible for their decision-making.

The COVID-19 pandemic has changed the organization of care, prioritizing the emergency fight against the epidemic.

The French High Authority of Health (HAS) has recommended maintaining individual TPE sessions by videoconference or telephone, based on the usual stages of the educational process. Several working groups have looked into remote TPE and recommendations have been issued in the form of practical advice but without questioning the participants, who did not participate in the reflection. No consensus, including health authorities, has been reached on this subject.

At Necker Hospital, ETPs were carried out remotely, by videoconference. Understanding remote therapeutic education by videoconference through lived experience, by means of a one-hour interview, of the caregivers who deliver it and the parents of patients or the patients who receive it, will make it possible to better understand the effects of remote mode on therapeutic education sessions but also on professional practices and on participants.

The benefit will be twofold: for caregivers: to facilitate the deployment of this new educational offer. For patients and their carers: give priority access to TPE to families who are far from the healthcare system or to patients who are too fragile to travel and thus reduce inequalities and geographical barriers.

DETAILED DESCRIPTION:
Chronic disease onset, due to its lasting and progressive nature, generates significant personal, family and socio-professional disabilities and difficulties. This situation requires active participation on the part of the patient, who must adopt protective behaviors in order to live better as much as possible.

Therapeutic patient education (TPE) is one of the mechanisms that will make patients as competent as possible to manage illness and treatment by helping them to be autonomous and responsible for their decision-making.

The COVID-19 pandemic has changed the organization of care, prioritizing the emergency fight against the epidemic. The TPE programs were also impacted by the pandemic.The French High Authority of Health (HAS) has recommended maintaining individual TPE sessions by videoconference or telephone, based on the usual stages of the educational process, without however defining clear recommendations for remote TPE. Several working groups have looked into remote TPE and recommendations have been issued in the form of practical advice without questioning the participants, who did not participate in the reflection. No consensus, including health authorities, has been reached on this subject.

At Necker Hospital, ETPs were carried out remotely, by videoconference. This new way of providing training required upstream preparation, reflection on the content, the use of digital tools and their mastery on the part of participants and speakers. The purpose of this qualitative study is to understand remote therapeutic education by videoconference through lived experience, by means of a one-hour interview, of the caregivers who deliver it and the parents of patients or the patients who receive it. The interviews will make it possible to better understand the effects of distant mode on therapeutic education sessions on participants but also on professional's practices. The benefit will be twofold: for caregivers: to facilitate the deployment of this new educational offer. For patients and their carers: give priority access to TPE to families who are far from the healthcare system or to patients who are too fragile to travel and thus reduce inequalities and geographical barriers.

ELIGIBILITY:
Inclusion Criteria:

* Understanding of the French language (oral and written) for all participants.
* Information and non-opposition of the subjects and of holders of parental authority of minor subjects.
* Caregivers: any health professional practicing videoconferencing therapeutic education can be included without age limit, regardless of gender, profession exercised (medical or paramedical) or the program concerned as long as the program is authorized (or declared) to authorized by the Ile-de-France Regional Health Agency (ARS).
* Participants: depending on the age of the patients, parents can be the exclusive target of therapeutic education (especially for young patients) or be present with their child during the sessions. The participants are the beneficiaries of therapeutic education either:

  * Parents/caregivers who have taken part in a videoconferencing TPE session (individual or collective) as part of a program authorized by the Ile-de-France ARS, regardless of their age, sex or the pathology concerned in the education program.
  * Patients: from 10 years old and only if the videoconferencing therapeutic education session was intended for them, regardless of gender or pathology.

Exclusion Criteria:

* Lack of training (40 hours) in TPE for caregivers.
* ETP program not authorized or not declared to the Ile-de-France ARS.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Caregivers and participants practicing/have beneficiating of videoconferencing therapeutic education at Necker-Enfants Malades hospital.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Understanding of remote therapeutic education by videoconference | 18 months
  Exploratory qualitative research of the lived experience of remote therapeutic education sessions by videoconference (phenomena) by interviewing participants and caregivers. Verbatim analysis of interviews by phenomenological qualitative method : collection, organization, and interpretation of textual material derived from talk or conversation to understand the phenomena and its meaning. The purpose of this approach is to bring out the categories of the phenomenon studied, each category representing a dimension of the phenomenon studied.

SECONDARY OUTCOMES:
Identify the particularities of distance therapeutic education and its success factors | 18 months
  Exploratory qualitative research of the lived experience of remote therapeutic education sessions by videoconference of participants and caregivers. Verbatim analysis of all the interviews, by the semio pragmatic phenomenology method, for identification of recurrences of theme to constitute a referencing of brakes and levers.
Develop recommendations levers for videoconferencing therapeutic education | 24 months
  From the synthesis of all the data analyzed (verbatim interview analysed with semio pragmatic phenomelogy method, by answering the question : what will you advice a person who will provide remote therapeutic education ?) collect a framework of recommendations (practices from the field) to carry out a remote therapeutic education session intended for caregivers and taking into account the expectations and needs of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Godot, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Radhia Dahmane, Study Director — Assistance Publique - Hôpitaux de Paris; Théo TENG, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No